CLINICAL TRIAL: NCT03869151
Title: The Impact of Pretreatment Lymphocyte to Monocyte Ratio on Clinical Outcome for Patient With HCC
Brief Title: Pretreatment Lymphocyte Monocyte Ratio on Outcome HCC Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Amany Aboalenen Amin (Other)
Responsible Party: Sponsor-Investigator, Amany Aboalenen Amin, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 17200000
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBC — lymphocyte and monocyte count

SUMMARY:
To assess the prognostic role of pretreatment LMR in hepatocellular carcinoma(HCC).

DETAILED DESCRIPTION:
The exact molecular mechanisms responsible for the prognostic impact of lymphocyte monocyte ratio in Heatocellular carcinoma are unclear.It has been suggested that cross-talk between the inflammatory response and tumor progression play a critical role in the initiation and progression of Heatocellular carcinoma. In the tumor microenvironment, inflammatory infiltrates have a large influence on the biological behavior of Heatocellular carcinoma.

Tumor-infiltrating lymphocytes, as representative component of the immune microenvironment ,are implicated in several stages of Heatocellular carcinoma progression, and Tumor-infiltrating lymphocytes phenotypes may be a predictor for favorable prognosis.

Conversely, low lymphocyte counts might result in an insufficient immunological reaction, which lead to inferior survival in multiple cancers.

Monocytes infiltrating tumor tissue are also involved in Heatocellular carcinoma development and progression. Activated monocytes in Heatocellular carcinoma micro environments can trigger and polarize T-cell responses and facilitate inflammation-induced tumor development.

Tumor-associated macrophages are derived from circulating monocytes. Tumor-associated macrophages can accelerate Heatocellular carcinoma cell proliferation,tumor-associated angiogenesis, and metastasis. Several studies showed that high infiltration of Tumor-associated macrophages predicted decreased survival in various cancers.

ELIGIBILITY:
Inclusion Criteria:

Patients with child A Hepatocellular carcinoma.

Exclusion Criteria:

* Patients with child C Hepatocellular carcinoma.
* Patients with heart failure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma patients
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2019-04-05 (Estimated); Primary Completion 2020-03-05 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
increased over all survival | 1 year
  Elevated pretreatment lymphocyte monocyte ratio may be a favorable prognostic factor for clinical outcomes in patients with hepatocellular carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: taha mahran, MD, Study Chair — Assiut University; ola abdelfatah, MD, Study Chair — Assiut University; aml ebraheem, MD, Study Director — Assiut University; amany amin, master, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided